CLINICAL TRIAL: NCT02709213
Title: Colitis Prospective Cohort Study: Determining the Aetiologies of Acute Colitis and Developing a Diagnostic Score to Identify Patients Requiring Specific Investigations
Brief Title: Determination of the Aetiologies of Acute Colitis and Early Identification of Patients Requiring Diagnostic Colonoscopy
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Principal Investigator, Jeremy Meyer, MD-PhD, University Hospital, Geneva
Other Study IDs: 14-211
Record Dates: First submitted 2016-03-02; First posted 2016-03-16 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Colitis
Keywords: Inflammatory chronic bowel disease; ICBD; Colorectal cancer; Infectious colitis
MeSH Terms: conditions — Colitis; Colorectal Neoplasms | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stools
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with CT-diagnosed acute colitis: Patients with symptomatic colitis (fever and/or pain and/or diarrhea) proven by computed tomography
  Interventions: Diagnostic Test: Diagnostic

INTERVENTIONS:
Diagnostic Test: Diagnostic — Determination of pathogens and faecal calprotectin in the stools
  Other Names: Stools: Faecal calprotectin; Stools: FilmArray GI panel (PCR multi-array)

SUMMARY:
The aetiologies of computed tomography-diagnosed acute colitis remain surprisingly unknown. Moreover, no diagnostic tool or clinical score allow to quickly determine or at least stratify the exact cause of colitis in patients admitted at an Emergency Ward and to direct them to the appropriate therapeutic care. The aims of the present study are to describe the presentation and aetiologies of acute colitis, and to develop diagnostic methods to guide patients admitted for acute colitis to the appropriate therapeutic care, notably colonoscopy.

DETAILED DESCRIPTION:
Colitis is the generic term that refers to an inflammation of a segment of the colonic tract confirmed by computed tomography. This pathology represents approximately 100-150 admissions per year in the Division of Digestive Surgery of the University Hospitals of Geneva.

The aetiologies of colitis are numerous and include all pathologies having the ability to cause the inflammation and thickening of the colon wall. Colites are classified according to their aetiologies into: infectious colitis (bacterial, parasitic or viral), inflammatory chronic bowel diseases (ulcerative colitis, Crohn's disease, others), ischaemic colitis and iatrogenic colitis (non-steroidal anti-inflammatory drugs, others). The aetiologies of colitis affect therapeutic care, since patients with infectious colitis will improve with appropriate antibiotics, those with inflammatory chronic bowel disease will require the introduction of an immunosuppressive therapy, and those with ischaemic colitis will only need a supportive treatment and a careful evaluation to detect any progression to bowel perforation that would prompt for surgery.

Therefore, numerous investigations are performed to determine the precise aetiology of colitis.

At the University Hospitals of Geneva, as well as in other centres, a microbiological analysis of faeces (routine PCR assay looking for Shigella spp., Salmonella spp. and Campylobacter spp.; PCR for Clostridium difficile as well as cultures for Vibrio spp. and Yersinia spp. (in option)) are performed in first intention. If these assays yield to the absence of a potential pathogen, a colonoscopy is performed to look for: 1) a tumour, 2) a chronic inflammatory bowel disease or 3) an ischaemic colitis. Patients in whom no aetiology can be found to explain the colonic inflammation are given a diagnosis of undetermined colitis.

However, the respective prevalences of the different aetiologies of colitis remain surprisingly unknown. Similarly, no diagnostic tool or clinical score allow to quickly determine or at least stratify the exact cause of colitis in patients admitted in the Emergency Ward and to direct them to the appropriate therapeutic care. As a consequence, all patients admitted with a diagnosis of computed tomography-proven colitis are subjected to broad-spectrum antibiotics associated with a 5-10 days hospitalisation for monitoring and investigations. Patients with negative microbiological examination of the stools will benefit from an early colonoscopy, a procedure that carries significant risks of complications and generates high costs. Moreover, the difficulties in the early identification of patients requiring endoscopy for suspected inflammatory chronic bowel disease or cancer may delay or even contribute to miss these diagnoses, especially if the acute phase of inflammatory chronic bowel disease has passed.

Considering the lack of evidences regarding the therapeutic care of colitis, we plan to constitute a cohort of 200 patients admitted for a first episode of computed tomography-proven colitis at the University Hospitals of Geneva. We will collect data related to 1) the history, clinical and para-clinical presentations at admission, 2) the results of the aetiological investigations; and we will complete the investigations by performing 3) a detailed microbiological examination of the stools using an accurate and rapid multi-array PCR assay (FilmArray, Biofire Diagnostics, Salt Lake City, USA), as well as 4) a dosage of faecal calprotectin (a marker of bowel inflammation).

The aims of the present study are to describe the presentation and aetiologies of colitis, and to develop diagnostic methods to guide patients admitted for acute colitis to the appropriate therapeutic care, with the objective to generate savings by shortening hospital stays and by better prescribing additional tests, including colonoscopy. We therefore think that an adequate and early patient stratification has important medical and economical values in this setting.

We expect: 1) to diagnose a higher proportion of infectious colitis than currently reported, and this within a shorter turnaround time, a finding that could serve as a basis to discuss and implement a reduction in the rate of colonoscopies, 2) to identify predicting factors, including faecal calprotectin, which would help distinguishing patients who require an endoscopic evaluation from others, among patients with negative microbiological examination of the stools.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 year old
* French speaking
* Informed consent
* ≥1 symptom compatible with an acute colitis (fever≥38°C ± acute abdominal pain ± diarrhoea) + colon wall thickening at computed tomography

Exclusion Criteria:

* Another diagnostic evoked by the radiologist (diverticulitis, tumor, ...)
* Patient with a positive history for: chronic inflammatory bowel disease ± colorectal cancer ± immunosuppression ± abdominal ascites
* Refusal of investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted at the Emergency Department with a first diagnosis of computed tomography-diagnosed acute colitis
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Determination of the aetiologies of colitis using microbiological examination of the stools +/- colonoscopy | <24 hours
  Determination of the aetiologies of colitis and classification into one of the following categories (in %): infectious colitis (bacterial, parasitic or viral), chronic inflammatory bowel diseases (ulcerative colitis, Crohn's disease, other), ischemic colitis and iatrogenic colitis (non-steroidal anti-inflammatory drugs, other). In first intention, the routine microbiological examination of the stools usually performed (PCR assay looking for Shigella spp., Salmonella spp. and Campylobacter spp.; PCR for Clostridium difficile as well as cultures for Vibrio spp. and Yersinia spp. (in option)) will be completed with a high-sensitivity multi-array PCR assay (FilmArray). If the routine microbiological examination of the stools yields to the absence of a potential pathogen, a colonoscopy will be performed to look for: 1) a tumour, 2) a chronic inflammatory bowel disease, or 3) an ischaemic colitis. Patients in whom no aetiology can be found will be given a diagnosis of indeterminate colitis.

SECONDARY OUTCOMES:
Identification of anamnestic, clinical and biological predicting factors for patients requiring diagnostic colonoscopy | <24 hours and at 1 year
  Variables related to patients presentation at admission will be detailed and collected, regarding anamnesis, clinical examination and para-clinical exams. Results of the investigations performed during hospitalization will be collected (microbiological examination of the stools, colonoscopy). Faecal calprotectin will be determined for all stool samples. The Geneva Tumour Registry will be searched for the occurrence of tumour at the site of colitis at 1 year after the initial diagnosis. Predictors of "positive" colonoscopy (inflammatory bowel disease, cancer) will be identified using univariate and multivariate logistic regression, analysing variables collected at admission and faecal calprotectin.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Meyer, MD-PhD, Principal Investigator — University Hospitals of Geneva, Switzerland
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No